CLINICAL TRIAL: NCT02953756
Title: Cognitive Outcome After Gamma Knife Radiosurgery in Patients With 1-10 Brain Metastases
Brief Title: Cognitive Outcome After Gamma Knife Radiosurgery in Patients With Brain Metastases (CAR-Study A)
Status: Completed | Type: Observational
Sponsor: Elisabeth-TweeSteden Ziekenhuis (Other)
Collaborators: Tilburg University (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Other Study IDs: 842003008
Record Dates: First submitted 2016-10-27; First posted 2016-11-03 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2020-02

CONDITIONS: Neoplasm Metastases
Keywords: Brain metastases; Cognition; Radiosurgery; Stereotactic radiosurgery; Gamma Knife Radiosurgery; Quality of Life; Fatigue; Anxiety; Depression
MeSH Terms: conditions — Neoplasm Metastasis; Brain Neoplasms; Fatigue; Anxiety Disorders; Depression | interventions — Radiosurgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stereotactic radiosurgery (SRS): Gamma Knife radiosurgery (GKRS)
  Interventions: Radiation: Gamma Knife radiosurgery

INTERVENTIONS:
Radiation: Gamma Knife radiosurgery — Gamma Knife radiosurgery will be performed with a Leksell Gamma Knife® Icon, Elekta Instruments, AB. Depending upon the tumor volume, a dose of 18-25 Gy will be prescribed with 99-100% coverage of the target

SUMMARY:
Stereotactic radiosurgery (SRS) is increasingly applied in patients with brain metastases (BM) and is expected to have less adverse effects on cognitive functioning than Whole Brain Radiation Therapy (WBRT). Because cognitive functions are essential for daily functioning, and may affect therapy compliance and quality of life in general, a full understanding of cognitive functioning in patients with BM after SRS is essential.

CAR-Study A is a prospective study to evaluate cognitive functioning in patients with 1-10 BM accepted for treatment with Gamma Knife radiosurgery (GKRS).

DETAILED DESCRIPTION:
CAR-Study A is a prospective study to evaluate cognitive functioning after GKRS in patients with 1-10 newly diagnosed brain metastases on a triple dose gadolinium-enhanced MRI-scan. Neuropsychological assessment will be performed at baseline and at 3, 6, 9, 12, 15, and 21 months after treatment. Follow-up assessments will be combined with 3-monthly MRI-scans.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven malignant cancer
* 1-10 newly diagnosed brain metastases on a triple dose gadolinium-enhanced MRI-scan
* Maximum total tumor volume 30 cm3
* Lesion ≥ 3 mm from the optic apparatus
* Age ≥ 18 years
* Karnofsky Performance Status (KPS) ≥ 70
* Anticipated survival > 3 months

Exclusion Criteria:

* No prior histologic confirmation of malignancy
* Primary brain tumor
* A second active primary tumor
* Small cell lung cancer
* Lymphoma
* Leukemia
* Meningeal disease
* Progressive, symptomatic systemic disease without further treatment options
* Prior brain radiation
* Prior surgical resection of brain metastases
* Additional history of a significant neurological or psychiatric disorder
* Participation in a concurrent study in which neuropsychological testing and/or health-related QOL assessments are involved
* Contra indications to MRI or gadolinium contrast
* Underlying medical condition precluding adequate follow-up
* Lack of basic proficiency in Dutch
* IQ below 85
* Severe aphasia
* Paralysis grade 0-3 according to MRC scale (Medical Research Council)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with 1-10 newly diagnosed brain metastases on a triple dose gadolinium-enhanced MRI-scan accepted for treatment with GKRS at the Gamma Knife Center Tilburg, The Netherlands.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2015-10; Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Change in verbal memory | Baseline and 3, 6, 9, 12, 15, and 21 months post GKRS
  Verbal memory is measured with the Hopkins Verbal Learning Test-Revised (HVLT-R)
Change in cognitive flexibility | Baseline and 3, 6, 9, 12, 15, and 21 months post GKRS
  Cognitive flexibility is measured with the Trail Making Test B (TMT B)
Change in word fluency | Baseline and 3, 6, 9, 12, 15, and 21 months post GKRS
  Word Fluency is measured with the Controlled Oral Word Association (COWA)
Change in working memory | Baseline and 3, 6, 9, 12, 15, and 21 months post GKRS
  Working memory is measured with the Wechsler Adult Intelligence Scale - Digit Span
Change in processing speed | Baseline and 3, 6, 9, 12, 15, and 21 months post GKRS
  Processing speed is measured with the Wechsler Adult Intelligence Scale - Digit Symbol
Change in motor dexterity | Baseline and 3, 6, 9, 12, 15, and 21 months post GKRS
  Motor dexterity is measured with the Grooved Pegboard (GP)

SECONDARY OUTCOMES:
Health Related Quality Of Life (HRQOL) | Baseline and 3, 6, 9, 12, 15, and 21 months post GKRS
  The Functional Assessment of Cancer Therapy-Brain (FACT-Br) is used to measure HRQOL.
Fatigue | Baseline and 3, 6, 9, 12, 15, and 21 months post GKRS
  Fatigue is measured with the Multidimensional Fatigue Inventory (MFI).
Depression and anxiety | Baseline and 3, 6, 9, 12, 15, and 21 months post GKRS.
  Depression and anxiety are measured with the Hospital Anxiety and Depression Scale (HADS).
Median Overall Survival | 12 months after GKRS
  Overall survival is defined as the time in months from the start of GKRS to the date of death or last contact if alive. Kaplan-Meier methods are used to estimate overall survival.
Local tumor control | 12 months after GKRS
  Local brain tumor control of the initial GKRS-treated lesions is defined as a complete, partial, or stable response, or less than a 25% increase in diameter on contrast-enhanced MRI follow-up and not requiring resection. Any initial treated lesions increased by more than 25% in diameter on contrast-enhanced MRI or required resection will be considered a local failure.
Distant tumor control | 12 months after GKRS
  Distant brain tumor control is defined as the absence of any new brain metastases, distinct from the initial GKRS-treated lesion(s), on follow-up MRI. The appearance of one or more new lesions in the brain by contrast-enhanced follow-up MRI is considered distant failure.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick EJ Hanssens, MD, Principal Investigator — Gamma Knife Center Tilburg, Elisabeth-TweeSteden Hospital, The Netherlands
Locations (1):
- Gamma Knife Center Tilburg, Elisabeth-TweeSteden Hospital, Tilburg, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Verhaak E, Schimmel WCM, Sitskoorn MM, Hanssens PEJ, Butterbrod E, Gehring K. The long-term course and relationship with survival of multidimensional fatigue in patients with brain metastases after Gamma Knife radiosurgery. J Cancer Res Clin Oncol. 2023 Sep;149(12):9891-9901. doi: 10.1007/s00432-023-04857-1. Epub 2023 May 30. PMID 37249646
- [Derived] Verhaak E, Schimmel WCM, Gehring K, Emons WHM, Hanssens PEJ, Sitskoorn MM. Health-related quality of life after Gamma Knife radiosurgery in patients with 1-10 brain metastases. J Cancer Res Clin Oncol. 2021 Apr;147(4):1157-1167. doi: 10.1007/s00432-020-03400-w. Epub 2020 Oct 6. PMID 33025282
- [Derived] Schimmel WCM, Gehring K, Hanssens PEJ, Sitskoorn MM. Cognitive functioning and predictors thereof in patients with 1-10 brain metastases selected for stereotactic radiosurgery. J Neurooncol. 2019 Nov;145(2):265-276. doi: 10.1007/s11060-019-03292-y. Epub 2019 Sep 24. PMID 31552588
- [Derived] Butterbrod E, Bruijn J, Braaksma MM, Rutten GM, Tijssen CC, Hanse MCJ, Sitskoorn MM, Gehring K. Predicting disease progression in high-grade glioma with neuropsychological parameters: the value of personalized longitudinal assessment. J Neurooncol. 2019 Sep;144(3):511-518. doi: 10.1007/s11060-019-03249-1. Epub 2019 Jul 24. PMID 31342318